CLINICAL TRIAL: NCT06352996
Title: Three-Dimensional Assessment of Maxillary Canine Retraction With and Without Power Arm: A Split-Mouth Randomized Controlled Trial
Brief Title: Three-Dimensional Assessment of Maxillary Canine Retraction With and Without Power Arm
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Anas Kassas, Dentist Anas Kassas, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Dentist Anas Kassas
Record Dates: First submitted 2024-03-28; First posted 2024-04-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Power Arm Canine Retraction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- power arm canine retraction (Experimental)
  Interventions: Other: Three-Dimensional Assessment of Maxillary Canine Retraction with Power Arm
- canine retraction without power arm (Experimental)
  Interventions: Other: Three-Dimensional Assessment of Maxillary Canine Retraction without Power Arm

INTERVENTIONS:
Other: Three-Dimensional Assessment of Maxillary Canine Retraction with Power Arm — A nickel titanium closed coil spring will be stretched from the mini-implant to the power arm will be used for canine retraction.
  Arms: power arm canine retraction
Other: Three-Dimensional Assessment of Maxillary Canine Retraction without Power Arm — A nickel titanium closed coil spring will be stretched from the mini-implant to the canine bracket will be used for canine retraction.
  Arms: canine retraction without power arm

SUMMARY:
Aim of the study: This trial will be conducted for three-dimensional assessment of canine retraction with and without power arm.

Materials and methods:Twenty patients with age range between 14 to 25 years. Before bonding, a hook will be attached to the canine bracket in one side only. Leveling and alignment then The first premolars will be extracted and mini-implant will be inserted.

Canine retraction using nickel titanium closed coil spring will start in the same day of upper first premolar extraction.

DETAILED DESCRIPTION:
Aim of the study: This trial will be conducted for three-dimensional assessment of canine retraction with and without power arm.

Participant and eligibility criteria:

Twenty patients will be recruited from the Department of Orthodontics at Mansoura University Pre-treatment records will be taken including: Intraoral and extraoral photographs, panoramic radiographs, cephalometric radiographs, and study models.

Intervention:

Written and informed consents will be taken from the patients. All patients will start the treatment by bonding fixed appliance (preadjusted edgewise, 0.018-in. slot, Roth prescription). Before bonding, a hook will be attached to the canine bracket in one side only. Leveling and alignment will be performed until reaching 0.017×0.025-in. nickel titanium arch wire. After 4 weeks of using the 0.017×0.025 arch wire, canine retraction phase will be initiated on 0.016×0.022 stainless steel arch wire.

After leveling and alignment, mini-implants will be inserted interradicular between the upper second premolar and upper first molar on each side. The mini-implant will be ligated to upper second premolar for indirect anchorage. The first premolars will be extracted at the same day of mini-implant placement.

Canine retraction will start in the same day of upper first premolar extraction. A nickel titanium closed coil spring will be stretched from the mini-implant to the power arm on one side, while direct retraction from the bracket will be used on the contralateral side. The retraction force will be adjusted to 150g using force gauge.

ELIGIBILITY:
Inclusion Criteria:

* Class II div 1 patients with age range between 14 to 25 years
* patients indicated for maxillary first premolar extraction
* increased over jet
* mild or no crowding in maxilla
* no previous orthodontic treatment
* no history of periodontal disease or bone loss
* good oral hygiene
* no systemic disease
* absence of canine morphological abnormalities.

Exclusion Criteria:

* patients not indicated for maxillary first premolar extraction
* decreased or no over jet
* moderate or severe crowding in maxilla
* previous orthodontic treatment
* history of periodontal disease or bone loss
* bad oral hygiene
* systemic disease
* canine morphological abnormalities.

Ages: 14 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-06-09 (Actual); Primary Completion 2024-03-09 (Actual); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Canine tipping | 4 months
  Intraoral scanning for maxillary arch will be recorded every month for each patient; at T0 (Immediately before canine retraction), T1 (after 1 month), T2 (2 months), T3 (3 months) and T4 (4 months). The four obtained digital models from each patient will be separately superimposed on each other.
  The change in the mesiodistal crown angulation of the canine will be calculated at each time point.
Canine mobility | 4 months
  The Periotest device will be used to measure the mobility of the canine immediately before retraction and repeated monthly for 4 months.
Implant stability | 4 months
  The Periotest device will be used to measure the stability of the mini-implant immediately before retraction and repeated monthly for 4 months.
Pain assessment | 1 week
  Pain assessment will be recorded by the visual analog scale (VAS) form. The participants will be informed to accomplish a visual analog scale diary containing 4 different times: four hours, 24 hours, 72 hours, and one week, following the beginning of the canine retraction.
  The pain level was on the 10-cm (100-mm) visual analog scale forms, with 0 (minimum) denoting no pain, while 100 (maximum) denoting sever pain.
canine rotation | 4 months
  Intraoral scanning for maxillary arch will be recorded every month for each patient; at T0 (Immediately before canine retraction), T1 (after 1 month), T2 (2 months), T3 (3 months) and T4 (4 months). The four obtained digital models from each patient will be separately superimposed on each other.
  The change in rotation of the canine will be calculated at each time point.
canine retraction rate | 4 months
  Intraoral scanning for maxillary arch will be recorded every month for each patient; at T0 (Immediately before canine retraction), T1 (after 1 month), T2 (2 months), T3 (3 months) and T4 (4 months). The four obtained digital models from each patient will be separately superimposed on each other.
  The retraction rate will be analyzed monthly and the total amount of canine retraction rate will be measured from cusp tip of the canine T0 to the same point in T4 for both sides.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry Mansoura University, Al Mansurah, Egypt

REFERENCES:
- [Derived] Kassas AN, Kamel AM, Mohammad MH, Fouda MAE, Montasser MA. Three-dimensional assessment of mini-implant supported maxillary canine retraction with and without power arm in class II division 1 patients: A split-mouth randomized trial. Int Orthod. 2025 Dec;23(4):101030. doi: 10.1016/j.ortho.2025.101030. Epub 2025 May 30. PMID 40449366